CLINICAL TRIAL: NCT01290926
Title: Sorafenib Plus Capecitabine Efficacy Assessment in Patients With Advanced Pre-treated Colorectal Cancer
Acronym: SoMore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Erasme University Hospital (Other); INDC Entité Jolimontoise (Unknown); Centre Hospitalier Chretien (Other); Universiteit Antwerpen (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Hospital Ambroise Paré Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2010-023695-91
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer
Keywords: advanced chemorefractory colorectal cancer; sorafenib; capecitabine; FDG-PET; early metabolic response
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Capecitabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine & Sorafenib (Experimental): Sorafenib 200mg in the morning,400mg in the evening; escalation to 400mg twice daily after 1 cycle, Oral, Continuous dosing Capecitabine 850mg/m2 twice daily, Oral Days 1-14, weeks 1-2
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: chemotherapy — sorafenib 600mg/day capecitabine 1250 mg/m²/day
  Other Names: Xeloda; Nexavar

SUMMARY:
Prospective non-randomized phase II study assessing the activity of the Capecitabine-Sorafenib combination by estimating overall survival of the study population at a fixed time point (6 months) and, as an exploratory analysis the overall survival of metabolic responders versus non-responders.

DETAILED DESCRIPTION:
Treatment doses :

Sorafenib 200mg in the morning,400mg in the evening; escalation to 400mg twice daily after 1 cycle Capecitabine 850mg/m2 twice daily Oral Days 1-14, weeks 1-2

Fluoro-Deoxy Glucose Positron Emitting Tomography (FDG-PET)imaging at baseline and after 17-21 days while on therapy.

Sample size justification/statistical analysis

Sample size has been estimated in order to be able to test the null hypothesis that the overall survival rate at 6 months is less than 30%. This hypothesis will be tested using a binomial distribution. The study should be able to reject the null hypothesis, using a 1-sided test with α = 0.025, with a power of 90% in case of a true overall survival ≥ 50% (rate at 6 months). The sample size required is 66 eligible patients (to be followed for 6 months minimum). Analysis will be done on all registered patients using an ITT approach on all eligible patients.

A co-primary endpoint is to compare the overall survival of patients assessed as early PET responders and of patients assessed as early PET non responders (the clinicians will remain blinded for PET response assessment). For this primary analysis, patients who will undergo the second PET assessment will be eligible and time zero for measuring survival will be the date of this second PET examination. It is anticipated that 95% of the patients will be eligible for the analysis with a 50% expected rate of early PET non-responders (result obtained from an unpublished study conducted at Jules-Bordet Institute). With 66 patients registered, we anticipate then that 63 patients will be available for the co-primary endpoint. With 63 patients and our assumption that the HR for the comparison between the survival distributions will be around 0.385 (based on the previously mentioned unpublished study), we will need using a two-sided logrank test at the 2.5% level (2.5% chosen because of the existence of 2 co-primary endpoints), 54 events (power of 90%). With 63 patients and a follow-up after accrual of 1 year, we should reach this number of 54 events. However, to account for another possible 5% drop-out (patient's refusal for undergoing the second PET examination for instance), sample size should be increased to 70 eligible patients.

However, our estimation of 50% expected rate of early PET responders is coming from a prospective unicentric cohort of 38 patients undergoing chemotherapy for 1st line or 2nd line treatment of advanced colorectal cancer with a few of them having received biological agents together with chemotherapy. Our estimation may then not be reliable due to small sample size and different patients population. If this rate of early PET responders proves to be higher, we should be prepared to increase our sample size for targeting the same power of 90%. For instance, if the rate is 67% instead of 50%, the required number of events would be 62 in-stead of 54. If the rate is 75%, the number of events should be increased to 73. The number of patients would have then to be adapted according to the rate of evaluable patients for this PET objective and the rate of patients lost to follow-up. For reassessing the required numbers of events, we did not change our hypothesis of detecting, if true, a hazard ratio of 0.385 in favor of early PET responders.

We plan, during the course of accrual, to assess the rate of patients evaluable for the PET objective, of early PET responders and, if possible the rate of patients lost to follow-up in order to check whether we need to review our planned sample size. However, no interim analysis will be done on the primary endpoints.

Secondary endpoints are to estimate progression-free survival and objective response rate, and to describe the adverse reactions associated with the study regimen in the study population. Also, to determine the correlation of early metabolic response, as assessed by FDG-PET/CT immediately before the first and the second cycles of treatment with the study regimen, with overall survival, progression-free survival, and response rate, and to determine the correlation of growth modulation index (GMI), defined as the time to progression under the study regimen over the time to progression under the latest regimen administered to the patient, with overall survival and progression-free survival.

The study is designed as a single-arm phase II study, with all patients accrued in one stage. No early stopping rules will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed colorectal cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* All standard chemotherapy agents (fluoropyrimidines, irinotecan, and oxaliplatin) and monoclonal antibodies (bevacizumab, cetuximab, and panitumumab) are allowed as administered therapy before study entry. No more than two lines of treatment for metastatic or recurrent disease are allowed, except for patients with KRAS-wt tumors, for which third line with anti-EGFR agents is allowed.
* Age over 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status ≤ 1.
* Participants must have normal organ and marrow function as defined below:
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* total bilirubin within 2 × normal institutional limits
* AST/ALT/PAKL levels < 5 × institutional upper limit of normal
* creatinine within 2 × normal institutional limits or creatinine clearance > 35mL/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants may not be receiving any other experimental agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib or capecitabine.
* Bleeding diathesis, history of cardiovascular ischemic disease or cerebrovascular incident within the last six months, or major surgery within four weeks.
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because sorafenib and capecitabine are antitumor agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with sorafenib or capecitabine, breastfeeding should be discontinued if the mother is treated with sorafenib or capecitabine. These potential risks may also apply to other agents used in this study.
* Uncontrolled Diabetes
* FDG PET/CT negative lesions or non metabolically assessable lesions (to small <2cm) at the base line FDG PET/CT
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall survival at 6 months fixed endpoint | 6 months
  The 2 primary co-endpoints are :
  1. To obtain a preliminary assessment about the activity of the combination by estimating overall survival of the study population at a fixed time point (6 months)
  2. To compare as an exploratory analysis the overall survival of metabolic responders versus non-responders.

SECONDARY OUTCOMES:
To estimate the Progression Free Survival (PFS) distribution of the study population | 12 months
To determine the objective response rate of the study population as assessed by standard imaging | 12 months
To describe the adverse reactions associated with the study regimen in the study population. | 12 months
To determine the correlation of early metabolic response, as assessed by FDG-PET/CT immediately before the first and the second cycles of treatment with the study regimen, with overall survival, progression-free survival, and response. | 12 months
To determine the correlation of growth modulation index (GMI), defined as the time to progression under the study regimen over the time to progression un-der the latest prior regimen administered to the patient, with overall survival and progression-free | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Principal Investigator — Jules Bordet Institute
Locations (7):
- Belgium (7):
  - Universiteit Ziekenhuis Antwerpen, Antwerp, Antwerpen
  - Cliniques Universitaires Saint Luc, Woluwe-Saint-Lambert, Brussels Capital
  - Institut Jules Bordet, Brussels
  - Hopital Erasme, Brussels
  - Entité Jolimontoise, La Louvière
  - Hopitaux St Joseph, Liège
  - CHU Ambroise Paré, Mons

REFERENCES:
- [Derived] Charette N, Vandeputte C, Ameye L, Bogaert CV, Krygier J, Guiot T, Deleporte A, Delaunoit T, Geboes K, Van Laethem JL, Peeters M, Demolin G, Holbrechts S, Flamen P, Paesmans M, Hendlisz A. Prognostic value of adipose tissue and muscle mass in advanced colorectal cancer: a post hoc analysis of two non-randomized phase II trials. BMC Cancer. 2019 Feb 12;19(1):134. doi: 10.1186/s12885-019-5319-8. PMID 30744591
- [Derived] Hendlisz A, Deleporte A, Delaunoit T, Marechal R, Peeters M, Holbrechts S, Van den Eynde M, Houbiers G, Filleul B, Van Laethem JL, Ceyssens S, Barbuto AM, Lhommel R, Demolin G, Garcia C, El Mansy H, Ameye L, Moreau M, Guiot T, Paesmans M, Piccart M, Flamen P. The Prognostic Significance of Metabolic Response Heterogeneity in Metastatic Colorectal Cancer. PLoS One. 2015 Sep 30;10(9):e0138341. doi: 10.1371/journal.pone.0138341. eCollection 2015. PMID 26421426